CLINICAL TRIAL: NCT01316185
Title: An Open Label, Dose-ranging Proof-of-concept Study Assessing the Safety and Efficacy of EBP921 in Therapy-naive Patients Chronically Infected With Delta Hepatitis (HDV)
Brief Title: Proof-of-concept Study Evaluating the Safety and Efficacy of EBP921 in Delta Hepatitis (HDV)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: the enrollment was slow and never completed.
Sponsor: Eiger BioPharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EBP-HDV 01-921-01
Record Dates: First submitted 2011-03-14; First posted 2011-03-16 (Estimated); Last update posted 2016-08-08 (Estimated); Status verified 2016-08

CONDITIONS: Hepatitis D
Keywords: Hepatitis D; HDV; Hepatitis
MeSH Terms: conditions — Hepatitis D; Hepatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): Low Dose for 28 days: n=4
  Interventions: Drug: EBP921
- Group 2 (Experimental): High Dose for 28 days; n=4
  Interventions: Drug: EBP921

INTERVENTIONS:
Drug: EBP921 — Patients randomized to receive low or high dose. All dosing of EBP921 should be taken with food.

SUMMARY:
The purpose of this study is to assess the optimal dose of EBP921 by comparing the efficacy and safety of 2 dose regimens in patients with chronic HDV.

DETAILED DESCRIPTION:
This is an open-label, phase 1b, proof-of-concept study to assess the safety and efficacy of EBP921, a prenylation inhibitor, in subjects chronically infected with delta hepatitis. Subjects will be randomized to receive one of two different doses of EBP921. Dosing will occur over 28-days and during that time, evidence of antiviral response will be assessed by frequent measurements of HDV-RNA via PCR assay. In addition, safety lab data will also be collected along with surveillance monitoring of HBV activity.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women age 18 or older with the capacity to give written informed consent
2. Patients with compensated chronic HDV infection as indicated by presence of anti-HDV in serum.
3. Liver biopsy should be performed within one-year of study screening and graded using the Knodell scoring system.
4. Presence of HDV antigen in liver tissue or HDV-RNA in serum.
5. Active HBV replication will not exclude patients.
6. Previous therapy with standard alpha-interferon or peginterferon will not exclude patients.
7. Patients who are HBV therapy-naïve or who previously received HBV antiviral therapy will be eligible. Patients currently taking HBV antiviral therapy will e considered on a case basis.
8. Female subjects of reproductive potential and female partners of male subjects should be on two reliable forms of contraception from the start of the study until 60 days from the end of EBP921 dosing.

Exclusion Criteria:

1. Severe neuropsychiatric disorders
2. History or clinical manifestations of significant metabolic, hematological, pulmonary, ischemic heart disease, significant or unstable heart disease, gastrointestinal, neurological, renal, urological, endocrine, ophthalmologic disorders including severe retinopathy, or immune-mediated disease
3. Pregnant or breast-feeding patients or the inability to practice adequate contraception during the conduct of the study
4. Underlying autoimmune/immune-deficiency disease (e.g., lupus, sarcoidosis, celiac disease, HIV antibody positive, AIDS)
5. Chronic (> 4 weeks duration) diarrhea
6. Body weight > 128 kg and < 40 kg
7. Uncompensated cirrhosis
8. Absolute neutrophil count less than 1500 per cubic millimeter
9. Platelet count less than 90,000 per cubic millimeter
10. Evidence of concurrent HCV infection with positive serum HCVRNA
11. Evidence of hepatocellular carcinoma
12. Active substance abuse (alcohol, inhaled or injected drugs) within the past 12 months
13. Diagnosis of malignancy in the previous five years excluding superficial dermatologic malignancies
14. Any experimental therapy in the previous 6 months prior to enrollment.

16. Patients with a history of multiple drug resistant HBV 17. Patients receiving interferon therapy for any reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2011-01; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Change in HDV-RNA | 28 days
  The primary efficacy endpoint will be the median change in HDV-RNA from baseline to HDV RNA nadir as measured by quantitative PCR during the 28-day dosing period.

SECONDARY OUTCOMES:
Change in HDV RNA from baseline to Day 7, 14, 28 and post therapy weeks 1,2,4,8 | 8 Weeks
  The median change in HDV RNA from baseline to Days 7, 14, 28, and post-therapy Weeks 1, 2, 4, and 8 of the study; the proportion of patients with alanine aminotransferase (ALT) normalization defined as ALT ≤ upper limit of normal for patients with ALT > ULN at baseline; assessment of peripheral blood mononuclear cell (PBMC) proliferation after 14 and 28 days exposure to EBP921; the percentage of patients with undetectable HDV RNA at Days 7, 14, 28, post-therapy Weeks 1, 2, 4, and 8; the median change in HBV DNA at Days 7, 14, 21, 28, 35, and 42, and HBsAg at Days 14, 28, and 42.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Murphy, MD, MPH, Study Director — Eiger BioPharmaceuticals, Inc.
Locations (2):
- United States (2):
  - San Francisco, California
  - Henry Ford Hospital, Detroit, Michigan